CLINICAL TRIAL: NCT03809637
Title: Phase II Study of Pemetrexed Plus Cisplatin in Patients With Refractory Soft Tissue Sarcoma
Brief Title: A Study of Pemetrexed Plus Cisplatin in Patients With Refractory Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0389
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pemetrexed+cisplatin (Experimental): Patients with metastatic sarcoma who underwent one chemotherapy regimens are treated with the combination of pemetrexed and cisplatin, and the treatment is repeated until the disease progression. pemetrexed 500 mg / m2 (day 1) and cisplatin 75 mg / m2 (day 1) are intravenously injected. 21 days is one cycle, and it is carried out by co-administration up to 6 cycles. After 7 cycles, intravenous injection of pemetrexed alone at intervals of 3 weeks until disease progression.
  Interventions: Drug: Pemetrexed, cisplatin

INTERVENTIONS:
Drug: Pemetrexed, cisplatin — Pemetrexed 500mg/m2, Intravenous, Q 3weeks. Cisplatin 75mg/m2, Intravenous, Q 3weeks. Combination administration : up to 6cycles After 6 cycle, pemetrexed alone is administered.

SUMMARY:
The yearly incidence of soft-tissue sarcomas(STS) in the USA is roughly 11,280 cases, and metastatic STS have a median overall survival of about 12 months. After the standard 1st line chemotherapy with doxorubicin, the only a few treatment option is available. Recently, pemetrexed, a novel multitargeted antifolate, has shown modest activity as a single agent lung cancer and mesothelioma. In patients with refractory STS, pemetrexed is well tolerated and moderately effective. Based on the background, investigators planned to conduct the phase II trial of pemetrexed in combination with cisplatin for metastatic/recurred soft-tissue sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced bone and soft tissue sarcoma with prior chemotherapy including anthracycline or ifosfamide
2. Measurable or evaluable disease (RECIST 1.1.)
3. Age ≥19 years
4. ECOG performance status of 0-2
5. Adequate laboratory findings

   * Absolute neutrophil count (ANC) ≥ 1500 /µL
   * Platelet count ≥ 75,000/ µL
   * Serum creatinine < 1.5 x upper limit of normal (ULN)
   * AST (SGOT) and ALT (SGPT) < 3 x upper limit of normal (ULN)
   * Total bilirubin <1.5 x upper limit of normal (ULN)
6. more than 3 months of expected survival
7. Provision of written informed consent prior to any study procedure

Exclusion Criteria:

1. Patient who has had chemotherapy, radiotherapy, or biological therapy within 2 weeks prior to entering the study'
2. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
3. Resectable lung metastases
4. Uncontrolled or active CNS metastasis and/or carcinomatous meningitis
5. Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma, thyroid cancer or cervical cancer in situ.
6. Uncontrolled medical conditions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
progression free rate | 12 weeks

SECONDARY OUTCOMES:
adverse event | every 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JH, Kim SH, Jeon MK, Kim JE, Kim KH, Yun KH, Jeung HC, Rha SY, Ahn JH, Kim HS. Pemetrexed plus cisplatin in patients with previously treated advanced sarcoma: a multicenter, single-arm, phase II trial. ESMO Open. 2021 Oct;6(5):100249. doi: 10.1016/j.esmoop.2021.100249. Epub 2021 Sep 2. PMID 34482181